CLINICAL TRIAL: NCT00519350
Title: Towards a High-fat Feeding Intervention Study: Identification of Markers for Inflammation and Organ Damage
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Jan-Willem Greve, University Hospital Maastricht
Other Study IDs: 074016
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2010-03

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis
Keywords: SIRS, sepsis and related syndromes
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- I: Liver surgery
  Interventions: Procedure: Blood collection
- II: Colon surgery
  Interventions: Procedure: Blood collection
- III: Femur Fracture
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — In arterial or venous lines already present, small amounts of blood will be collected at certain timepoints following operation

SUMMARY:
Patients undergoing major surgery, trauma or burns are prone to develop an exacerbated inflammatory response, which is potentially lethal to the individual. Recently, the researchers' group showed in a rodent model of hemorrhagic shock that high-fat feeding administered before shock attenuates inflammation and reduces intestinal and hepatic damage. In the mechanism that underlies this protective effect, the release of cholecystokinin in gut wall and activation of efferent vagus bundles are crucial events. Before investigating the effect of high-fat nutrition in clinical setting, suitable markers of inflammation and organ damage need to be selected. In this study, blood will be collected in patients undergoing different types of operations. Consequently several markers for inflammation and organ damage will be determined. Hence, suitable parameters for a future high-fat intervention study will be selected.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* elective liver / colon / femur surgery

Exclusion Criteria:

* Acute inflammation
* Chronic Obstructive Respiratory Disease
* Recent history of abdominal pain or diarrhea
* BMI < 18.5
* Alcohol or Drugs abuses
* Recent intake of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Maastricht University Hospital area undergoing one of selected types of surgery
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Greve, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands